CLINICAL TRIAL: NCT00097708
Title: A Double-Blind, Placebo Controlled Trial of an Experimental Medication For the Treatment of Generalized Anxiety Disorder
Brief Title: Experimental Medication For the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP 04-001-01
Record Dates: First submitted 2004-11-29; First posted 2004-11-30 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Anxiety Disorder
Keywords: Double Blind, Placebo controlled, Safety and Efficacy; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

INTERVENTIONS:
Drug: experimental anti-anxiety drug

SUMMARY:
The purpose of this study is to determine whether an experimental anti-anxiety medication is effective in the treatment of Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
Protocol 04-001-01

The primary objective of the study is to assess, under controlled conditions, the safety and efficacy of an experimental anti-anxiety medication relative to placebo in subjects with generalized anxiety disorder (GAD).

The secondary objective of the study is to study algorithms for discontinuation of an experimental anti-anxiety medication.

Recruiting: Participants are currently being recruited and enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 65 years of age will be eligible to participate if they satisfy the DSM-IV-TR criteria for the diagnosis of GAD.

Exclusion Criteria:

* No other primary psychiatric diagnosis besides GAD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2004-11; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Murray Stein, MD, Study Chair — University of California, San Diego
Locations (50):
- United States (50):
  - Birmingham Research Group, Inc., Birmingham, Alabama
  - Crest Clinical Trials, Inc., Anaheim, California
  - Southwesten Research, Inc., Beverly Hills, California
  - Southwestern Research Institute, Burbank, California
  - University of California - San Diego - Dept of Psychiatry, San Diego, California
  - Clinical Innovations, Santa Ana, California
  - Stanford University Medical Center, Stanford, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - New Britain General Hospital, New Britain, Connecticut
  - Florida Clinical Research Center, Bradenton, Florida
  - ACT Clinical Research, DeLand, Florida
  - University Clinical Research DeLand, Inc., DeLand, Florida
  - Sarkis Clinical Trials, Gainsville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - Institute of Research in Psychiatry, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Institute of Medicine and Research, Marietta, Georgia
  - Radiant Research, Boise, Idaho
  - American Medical Research, Inc., Oak Brook, Illinois
  - Peak Medical Research, LLC, Owensboro, Kentucky
  - New Orlean Medical Institute, Metairie, Louisiana
  - Brentwood Research Institute, Shreveport, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Pivotal Research Centers - Detroit, Royal Oak, Michigan
  - MedClin Research, St Louis, Missouri
  - CNS Research Institute (CRI), Clementon, New Jersey
  - ClinSearch, Inc., Kenilworth, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Laureate Psychiatric Clinic and Hospital, Tulsa, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Eugene, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - CNS Research Institute, Philadelphia, Pennsylvania
  - Southeast Health Consultants, LLC, Charleston, South Carolina
  - CNS, Inc., Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Research Across America, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Comprehensive Neuroscience of Northern Virginia, Falls Church, Virginia
  - Dominion Clinical Research, Inc., Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- OROS Alprazolam: OROS (osmotic [controlled] release oral [delivery] system) alprazolam administered orally once a day, titrated to maximum beneficial dose, 1,2,3,4,5, or 6 mg/day
- IR Alprazolam: IR (immediate release) alprazolam (Xanax) administered orally in divided dose (3 times daily), titrated to maximum beneficial dose, 1,2,3,4,5, or 6 mg/day
- Placebo: OROS (osmotic [controlled] release oral [delivery] system) placebo administered orally once a day.
Period: Overall Study
Arm/Group | OROS Alprazolam | IR Alprazolam | Placebo
Started | 173 | 176 | 162
Intent-to-Treat (ITT) | 165 | 169 | 149
Treated | 171 | 176 | 160
Completed | 109 | 120 | 97
Not Completed | 64 | 56 | 65

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OROS Alprazolam | IR Alprazolam | Placebo | Total
Number analyzed (Participants) | 165 | 169 | 149 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.00) | 38.9 (12.02) | 38.5 (11.13) | 38.8 (11.72)
Age, Customized [Number; unit: participants]
  < 40 years | 87 | 90 | 91 | 268
  40 - < 65 years | 76 | 78 | 58 | 212
  >=65 years | 2 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 113 | 103 | 311
  Male | 70 | 56 | 46 | 172
Region of Enrollment [Number; unit: participants]
  United States | 165 | 169 | 149 | 483

OUTCOME MEASURES:

1. Primary Outcome: Change in HAM-A Total Score
Description: Hamilton Anxiety Rating Scale (HAM-A). Each of 14 symptoms categories is rated from 0=not present to 4=very severe. Numbers for all categories are summed to produce the total score. Total score ranges from 0=anxiety symptoms not present to 56=very severe anxiety symptoms across all 14 categories.
Time Frame: Baseline to week 8
Measure: Least Squares Mean (Full Range); unit: Units on a Scale
Arm/Group | OROS Alprazolam | IR Alprazolam | Placebo
Number analyzed (Participants) | 162 | 159 | 145
Units on a Scale | -12.9 [-33 to 9] | -15.7 [-36 to 5] | -12.5 [-35 to 4]
Statistical Analysis 1: Comparison: OROS Alprazolam vs Placebo; Test type: Superiority or Other; p = 0.6540, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.2 to 1.4]
Statistical Analysis 2: Comparison: IR Alprazolam vs Placebo; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Net) = -3.2, 95% CI 2-sided [-5.0 to -1.4]
Statistical Analysis 3: Comparison: OROS Alprazolam vs IR Alprazolam; Test type: Superiority or Other; p = 0.0015, ANCOVA; Mean Difference (Net) = 2.8, 95% CI 2-sided [1.1 to 4.5]

ADVERSE EVENTS:
Arm/Group | OROS Alprazolam | IR Alprazolam | Placebo
Serious Adverse Events (participants affected / at risk) | 6/171 | 1/176 | 0/160
Other Adverse Events (participants affected / at risk) | 140/171 | 141/176 | 118/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OROS Alprazolam (N=171) | IR Alprazolam (N=176) | Placebo (N=160)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intentional Self-Injury (Psychiatric disorders) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OROS Alprazolam (N=171) | IR Alprazolam (N=176) | Placebo (N=160)
Nausea (Gastrointestinal disorders) | 13 | 17 | 19
Diarrhoea (Gastrointestinal disorders) | 9 | 15 | 12
Dry Mouth (Gastrointestinal disorders) | 6 | 9 | 11
Fatigue (General disorders) | 25 | 23 | 14
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 20 | 9
Somnolence (Nervous system disorders) | 48 | 47 | 11
Headache (Nervous system disorders) | 23 | 27 | 28
Dizziness (Nervous system disorders) | 19 | 29 | 10
Sedation (Nervous system disorders) | 13 | 18 | 6
Insomnia (Psychiatric disorders) | 11 | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other